CLINICAL TRIAL: NCT07271706
Title: The Effect of Laughter Yoga on Self-management and Comfort in Type 2 Diabetes Patients
Brief Title: The Effect of Laughter Yoga in Type 2 Diabetes Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Betül Bal, Lecturer Doctor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Yobu
Record Dates: First submitted 2025-11-21; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Diabetic; Laughter Yoga; Comfort
Keywords: laughter yoga; diabetic; comfort; self-governance
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Laughter Yoga Protocol
  The Laughter Yoga program administered to participants in the intervention group will be structured in accordance with protocols used in similar studies in the literature. The program will be conducted twice a week for four weeks. Each session will last approximately 40 minutes and will include the following four components:
  1. Warm-up and Breathing Exercises (5-7 minutes) Participants will engage in gentle warm-up movements and guided breathing exercises to promote relaxation, increase body awareness, and prepare for laughter activities.
  2. Laughter Exercises (15-20 minutes) Participants will perform voluntary laughter through instructor-guided techniques. These exercises are designed to activate the diaphragm, enhance oxygenation, stimulate positive emotional states, and increase parasympathetic activity. Techniques may include greeting laughter, clapping rhythms, playful interactions, and simulated laughter sequences.
  3. Diaphragmatic Breathing and Relaxat
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- Laughter yoga (Experimental)
  Interventions: Behavioral: Laughter yoga

INTERVENTIONS:
Behavioral: Laughter yoga — Arm Description: A structured laughter yoga program delivered twice weekly for four weeks. Each 40-minute session includes warm-up and breathing exercises (5-7 min), guided laughter exercises (15-20 min), diaphragmatic breathing and relaxation (5-7 min), and mindfulness-based closing practices (3-5 min). Conducted by a certified facilitator.
  Arms: Laughter yoga

SUMMARY:
The purpose of this study is to examine the effect of laughter yoga on self-management skills and comfort levels in patients with Type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes is a major global health problem affecting more than 537 million adults worldwide, a number expected to rise substantially in the coming decades. Type 2 diabetes, the most prevalent form, requires consistent self-management to maintain glycemic control and prevent complications. However, individuals living with chronic illness often experience ongoing physiological fatigue and emotional stress, which can reduce self-efficacy and hinder engagement in self-management behaviors. Comfort, identified as an important psychological resource, plays a supportive role in sustaining these behaviors.

Katharine Kolcaba's Comfort Theory proposes that health behaviors can be positively influenced by enhancing individuals' physical, psychospiritual, sociocultural, and environmental comfort. Laughter Yoga-a mind-body intervention combining intentional laughter with breathing and relaxation techniques-has been shown to reduce stress, improve mood, and increase parasympathetic activity. Previous studies involving individuals with Type 2 diabetes have reported reductions in HbA1c, decreased stress levels, and improved quality of life following Laughter Yoga interventions. However, limited research has simultaneously examined its effects on both self-management behaviors and comfort levels.

This study aims to evaluate the effects of Laughter Yoga on self-management behaviors and comfort levels among individuals with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Type 2 diabetes
* Age 18 years or older
* Willingness to participate in the Laughter Yoga intervention
* Ability to read and comprehend Turkish

Exclusion Criteria

* Diagnosis of Type 1 diabetes
* Participation in individual psychotherapy or group-based psychological intervention programs
* Experience of a recent loss within the past month (e.g., death, divorce)
* Presence of any psychiatric diagnosis
* Use of psychiatric medication
* Severe visual or hearing impairment preventing active participation in the intervention
* Pregnancy or breastfeeding
* Limitations in reading or comprehending Turkish

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Diabetes Self-Management Score (Diabetes Self-Management Questionnaire - DSMQ) | Baseline (Day 0) and Week 4
  The Diabetes Self-Management Questionnaire (DSMQ), originally developed by Schmitt et al. (2013), will be used to evaluate diabetes self-management behaviors. The DSMQ consists of 16 items and four subscales:
  Glucose Management
  Dietary Control
  Physical Activity
  Health-Care Use
  Items are rated on a 4-point Likert scale (0-3). Seven items are scored positively, and nine items are reverse-scored. Total scores are calculated by dividing the raw score by the maximum possible score and multiplying by 10. The resulting values range from 0 to 10, with higher scores indicating better diabetes self-management.
Comfort Level Score (General Comfort Questionnaire - Short Form) | Baseline (Day 0) and Week 4
  The General Comfort Questionnaire - Short Form, developed by Kolcaba (2006), will be used to assess comfort levels across physical, psychospiritual, environmental, and social domains. The scale consists of 28 items and three subscales:
  Relief
  Ease
  Transcendence
  Items are rated on a 6-point Likert scale (1-6). Negative items are reverse-scored. The total comfort score ranges from 1 to 6, with higher scores indicating greater comfort.